CLINICAL TRIAL: NCT07024953
Title: Setting the Agenda: A Pilot Stepped Wedge Cluster Randomized Trial of a Structured Clinical Visit Agenda-Setting Intervention for Rural-Residing People With Advanced Chronic Kidney Disease
Brief Title: The Agenda-Setting for Kidney Disease Trial
Acronym: ASK
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Dartmouth College (Other); University of Washington (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Catherine Hylas Saunders, Scientist & Assistant Professor of Medicine and of Health Policy & Clinical Practice, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY02002598_1; 1K01DK139400 (NIH)
Record Dates: First submitted 2025-06-09; First posted 2025-06-17 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Chronic Kidney Disease Stage 4; Chronic Kidney Disease Stage 5
Keywords: Chronic Kidney Disease; Chronic kidney disease stage 4; Chronic kidney disease stage 5; Agenda-setting; Rural; Patient engagement; Randomized trial; Participatory research
MeSH Terms: conditions — Renal Insufficiency, Chronic; Patient Participation

STUDY DESIGN:
Intervention Model Description: Stepped wedge randomized controlled trial with clustered cross-over assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 is Usual Care (No Intervention): The clinicians in the nephrology clinic will proceed with usual care without intervention from the study team.
- Arm 2 is Clinical Visit Agenda Setting Tool Intervention (Experimental): The study team will implement a structured clinical visit agenda-setting (SAS) intervention customized for advanced chronic kidney disease, called Chronic Kidney Disease (CKD) Topics.
  Interventions: Other: Chronic Kidney Disease Structured Agenda-Setting Tool

INTERVENTIONS:
Other: Chronic Kidney Disease Structured Agenda-Setting Tool — Chronic Kidney Disease (CKD) Topics is a novel clinical visit agenda-setting intervention developed through participatory research methods for people with CKD living in rural areas. CKD Topics includes structured discussion topic areas.
  Arms: Arm 2 is Clinical Visit Agenda Setting Tool Intervention

SUMMARY:
The goal of this clinical trial is to learn if a tool with a list of discussion topics, called a structured clinical visit agenda-setting intervention (SAS), works for people with advanced chronic kidney disease (CKD) who receive care at a clinic that serves people who live in rural areas. The SAS is called CKD Topics. The researchers will compare the SAS intervention to usual care (the way clinicians usually practice) to see how well it works for people with advanced CKD. This is a special type of clinical trial called a stepped wedge randomized clinical trial (RCT). In this type of trial, every participant will get to experience both usual care and CKD Topics, but for different amounts of time.

The researchers will learn if doing a clinical trial of CKD Topics is possible (feasible) and get information about how well CKD Topics helps people with advanced CKD shape visit discussions (self-advocacy) in their appointments with their clinicians. The information the researchers collect in this trial will help design a future trial with more participants.

The main questions the researchers aim to answer are:

* Is it possible to conduct this type of study of a SAS intervention? i.e. feasibility
* Does the SAS intervention help people with advanced CKD shape discussions (self-advocacy) with their clinicians? If so, how much? i.e. preliminary efficacy

DETAILED DESCRIPTION:
This stepped-wedge pilot randomized controlled trial (RCT) is to test a new structured agenda-setting (SAS), called the Chronic Kidney Disease (CKD) Topics Agenda-Setting Tool, with patients, their care partners and their clinicians. This is a pilot study, so the researchers are collecting feasibility data to determine if a larger, fully-powered RCT can be moved forward. The researchers are also collecting preliminary efficacy data, which will help the design of a future study on the efficacy of clinical visits for people with advanced CKD.

This study has two arms: 1) a usual care arm, and 2) an intervention arm where participants and their nephrology physicians will use CKD Topics during their visits. Physicians will initially be randomly assigned to one of three clusters, with two attending physicians and one fellow physician in each cluster. Each cluster will start out practicing usual care for at least eight months during the enrollment period. After that initial 8 months, one cluster will cross over to the intervention arm every four months, by using the CKD Topics tool in their visits, in what's called the rollout period. At 16 months into the trial, all clusters will be on the intervention arm, using CKD topics with patients, and will do so for the remaining 12 months of the trial.

Patient participants will be enrolled in the study arm to which their physicians have been randomized. Participation is expected to last 24 months for patients and clinicians, and participants may use CKD Topics more than once during the study period. The researchers expect 108 patient participants, and nine clinicians will enroll in the study. Every participant will receive a baseline survey after enrollment and four subsequent surveys.

The procedures in this study will include screening patients for study eligibility, consenting them to participate in study activities such as filling out surveys. The intervention, CKD topics, itself will be administered as quality improvement so will not be included as a research activity needing consent.

Future Directions: Findings from this trial will forecast a range of participants required in the sample for a full-scale RCT and illustrate "proof of concept" for a future trial which will evaluate the intervention's impact on patient self-advocacy and clinical care outcomes in rural CKD populations.

ELIGIBILITY:
Inclusion Criteria:

* Adults >18 years old who have been diagnosed with advanced CKD (stages 4-5).
* Care partners, clinicians and staff supporting these CKD patients who are willing and able to provide informed consent
* English-speaking
* Able to provide informed consent
* Patient must be attending outpatient visits *(in-person and/or telehealth allowable).

Exclusion Criteria:

* Children under 18 years old will not be included
* Non-English-speaking patients and/or care partners
* Patients on dialysis
* Individuals unable or unwilling to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2026-09-01 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Primary Feasibility Outcome | From enrollment to the end of treatment at 16 months
  The primary outcome will be feasibility, assessed by the proportion of patients who received the intervention.

SECONDARY OUTCOMES:
Secondary Feasibility Outcome | From enrollment to the end of treatment at 16 months
  The secondary outcome will be feasibility assessed by the clinicians' intention to continue the intervention use, measured in a survey.

OTHER OUTCOMES:
Primary Process Outcome: Enrollment Rate | From enrollment to the end of treatment at 16 months
  As measured by participant enrollment in Redcap.
Secondary Process Outcome: Loss to follow-up | From enrollment to the end of treatment at 16 months
  As measured by participant dropout (loss to follow-up) in Redcap.
Preliminary Efficacy Outcome: Patient Self-Advocacy Scale (PSAS) | From enrollment to the end of treatment at 16 months
  The Patient Self-Advocacy Scale (PSAS); a 12-item validated scale assessing the latent construct of perceived self-advocacy for patients.
Preliminary Efficacy Outcome: Patient self-efficacy | From enrollment to the end of treatment at 16 months
  Patient self-efficacy measured using the Ask, Understand, Remember Assessment, (AURA); a validated 4-item assessment of self-efficacy completed by patients.
Preliminary Efficacy Outcome: Patient self-management | From enrollment to the end of treatment at 16 months
  Patient demonstration of self-management using the Perceived Medical Condition Self-Management Scale; an 8-item instrument validated to assess self-management among CKD patients; correlated with treatment adherence.
Preliminary Efficacy Outcome: Unplanned hospitalization or emergency department visit | From enrollment to the end of treatment at 16 months
  Unplanned hospitalization or emergency department visit. EHR chart review and patient self-report.
Preliminary Efficacy Outcome: Serious Illness Experience | From enrollment to the end of treatment at 16 months
  Serious illness experience measured by the consideRATE questions; a validated 8-item, plain language (2nd grade) patient-reported experience measure (PREM) with Likert-like response options for patients, and care partners.
Preliminary Efficacy Outcome: Respect Experience Assessment | From enrollment to the end of treatment at 16 months
  Respect experience assessment measured by the "Heard and Understood" tool. Heard and Understood is a validated Single-item PREM with Likert-like response options for patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No
The study will use standard processing and documentation protocols adopted by the Inter-university Consortium for Political and Social Research (ICPSR) for data formats, dictionaries, variable names, descriptions, and labels. An XML schema using Data Documenting Initiative standards will also be used for codebooks and other metadata as appropriate. The researchers will share RCT process and outcomes data in CSV files via openICPSR, which is a self-publishing repository for social, behavioral and health science data and part of the ICPSR.

REFERENCES:
- [Background] Brashers DE, Haas SM, Neidig JL. The patient self-advocacy scale: measuring patient involvement in health care decision-making interactions. Health Commun. 1999;11(2):97-121. doi: 10.1207/s15327027hc1102_1. PMID 16370972
- [Background] Clayman ML, Pandit AU, Bergeron AR, Cameron KA, Ross E, Wolf MS. Ask, understand, remember: a brief measure of patient communication self-efficacy within clinical encounters. J Health Commun. 2010;15 Suppl 2(Suppl 2):72-9. doi: 10.1080/10810730.2010.500349. PMID 20845194
- [Background] Frankel RM, Salyers MP, Bonfils KA, Oles SK, Matthias MS. Agenda setting in psychiatric consultations: an exploratory study. Psychiatr Rehabil J. 2013 Sep;36(3):195-201. doi: 10.1037/prj0000004. Epub 2013 Jul 1. PMID 23815174
- [Background] Gramling R, Stanek S, Ladwig S, Gajary-Coots E, Cimino J, Anderson W, Norton SA; AAHPM Research Committee Writing Group; Aslakson RA, Ast K, Elk R, Garner KK, Gramling R, Grudzen C, Kamal AH, Lamba S, LeBlanc TW, Rhodes RL, Roeland E, Schulman-Green D, Unroe KT. Feeling Heard and Understood: A Patient-Reported Quality Measure for the Inpatient Palliative Care Setting. J Pain Symptom Manage. 2016 Feb;51(2):150-4. doi: 10.1016/j.jpainsymman.2015.10.018. Epub 2015 Nov 17. PMID 26596879
- [Background] Hemming K, Haines TP, Chilton PJ, Girling AJ, Lilford RJ. The stepped wedge cluster randomised trial: rationale, design, analysis, and reporting. BMJ. 2015 Feb 6;350:h391. doi: 10.1136/bmj.h391. No abstract available. PMID 25662947
- [Background] Makoul G, Krupat E, Chang CH. Measuring patient views of physician communication skills: development and testing of the Communication Assessment Tool. Patient Educ Couns. 2007 Aug;67(3):333-42. doi: 10.1016/j.pec.2007.05.005. Epub 2007 Jun 18. PMID 17574367
- [Background] Saunders CH, Durand MA, Kirkland KB, MacMartin MA, Barnato AE, Elwyn G. Psychometric assessment of the consideRATE questions, a new measure of serious illness experience, with an online simulation study. Patient Educ Couns. 2022 Jul;105(7):2581-2589. doi: 10.1016/j.pec.2022.01.002. Epub 2022 Jan 22. PMID 35260261
- [Background] Saunders CH, Durand MA, Scalia P, Kirkland KB, MacMartin MA, Barnato AE, Milne DW, Collison J, Bennett A, Wasp G, Nelson E, Elwyn G. "It helps us say what's important..." Developing Serious Illness Topics: A clinical visit agenda-setting tool. Patient Educ Couns. 2023 Aug;113:107764. doi: 10.1016/j.pec.2023.107764. Epub 2023 Apr 18. PMID 37150152
- [Background] Saunders CH, Durand MA, Scalia P, Kirkland KB, MacMartin MA, Barnato AE, Milne DW, Collison J, Jaggars A, Butt T, Wasp G, Nelson E, Elwyn G. User-Centered Design of the consideRATE Questions, a Measure of People's Experiences When They Are Seriously Ill. J Pain Symptom Manage. 2021 Mar;61(3):555-565.e5. doi: 10.1016/j.jpainsymman.2020.08.002. Epub 2020 Aug 16. PMID 32814165
- [Background] Sierpe A, Yen RW, Stevens G, Van Citters AD, Elwyn G, Saunders CH. Agenda-setting in the clinical encounter: A systematic review protocol. PLoS One. 2024 Oct 24;19(10):e0312613. doi: 10.1371/journal.pone.0312613. eCollection 2024. PMID 39446854
- [Background] Weiner BJ, Lewis CC, Stanick C, Powell BJ, Dorsey CN, Clary AS, Boynton MH, Halko H. Psychometric assessment of three newly developed implementation outcome measures. Implement Sci. 2017 Aug 29;12(1):108. doi: 10.1186/s13012-017-0635-3. PMID 28851459
- [Background] Wild MG, Wallston KA, Green JA, Beach LB, Umeukeje E, Wright Nunes JA, Ikizler TA, Steed J, Cavanaugh KL. The Perceived Medical Condition Self-Management Scale can be applied to patients with chronic kidney disease. Kidney Int. 2017 Oct;92(4):972-978. doi: 10.1016/j.kint.2017.03.018. Epub 2017 May 18. PMID 28528132